CLINICAL TRIAL: NCT01515475
Title: Glasses Versus Observation for Moderate Hyperopia in Young Children (HTS1)
Brief Title: Hyperopia Treatment Study 1 (HTS1) - Glasses vs Observation
Acronym: HTS1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: Pediatric Eye Disease Investigator Group (Network); National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HTS1; 2U10EY011751 (NIH)
Record Dates: First submitted 2012-01-11; First posted 2012-01-24 (Estimated); Results first posted 2019-05-09 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Hyperopia
Keywords: Hyperopia; Glasses
MeSH Terms: conditions — Hyperopia | interventions — Eyeglasses

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Glasses (Active Comparator): Glasses are prescribed at enrollment and worn per protocol throughout the duration of the study.
  Interventions: Procedure: Glasses
- Observation (Placebo Comparator): Glasses will not be prescribed unless the patient has confirmation of one or more deterioration criteria as described in the protocol.
  Interventions: Procedure: Glasses

INTERVENTIONS:
Procedure: Glasses — Glasses will be prescribed at enrollment with the sphere cut symmetrically by 1.00D and full cylinder correction.

SUMMARY:
The purpose of this study is to compare visual acuity outcomes and development of strabismus after a 3-year follow-up period in children age 12 to <72 months with moderate hyperopia (spherical equivalent +3.00D to +6.00D) who are prescribed glasses either immediately or only after confirmation of pre-specified deterioration criteria.

DETAILED DESCRIPTION:
Moderate and high hyperopia are associated with the development of strabismus and amblyopia. The primary aims of treatment for asymptomatic moderate and high hyperopia in preschool children are to facilitate the development of normal visual acuity and to prevent the development of esotropia and amblyopia. Treatment consists of optical correction, typically using glasses. For children with high hyperopia (>+5.00D) and without strabismus or amblyopia, there is general consensus that a correction should be prescribed. Nevertheless, for children with moderate hyperopia (+3.00D to +5.00D) without strabismus or amblyopia, there is less consensus among pediatric eye care professionals. A survey by Lyons et al found that for a 2-year-old child with hyperopia greater than +3.00D, 65% of optometrists would prescribe glasses compared to 25% of ophthalmologists; for a 4-year old with hyperopia greater than +3.00D, 67% of optometrists would prescribe compared with 42% of ophthalmologists. The American Association for Pediatric Ophthalmology and Strabismus (AAPOS) recommends correcting +4.00D or more in 2 to 7 year olds and the American Academy of Ophthalmology recommends a threshold of +4.50D for correction in 2-to 3-year olds. Unlike ophthalmology, optometry does not provide specific recommendations based on age and level of refractive error. Such variation in practice highlights the lack of rigorously collected scientific evidence for the management of this condition. Across all levels of hyperopia, most ophthalmologists and optometrists usually prescribe less than the full cycloplegic refraction (71% in the Lyons survey) when no strabismus or amblyopia is present.

The rationale for proactively correcting moderate hyperopia in an asymptomatic child is the prevention of esotropia, amblyopia, or asthenopia. The argument against correcting moderate hyperopia in an asymptomatic child is the expense and inconvenience of glasses that might be unnecessary and the potential disruption of emmetropization in infants and toddlers. At present, it remains uncertain whether correction of moderate hyperopia is beneficial in terms of visual acuity outcomes or strabismus development. There is some evidence that using partial correction of hyperopia allows emmetropization to take place.

If refractive correction of moderate hyperopia does not reduce the incidence of amblyopia and/or esotropia compared to no refractive correction, then glasses can be avoided. However, if correcting moderate hyperopia does reduce the development of amblyopia and/or esotropia, then the benefits of preemptive refractive correction will have been identified.

ELIGIBILITY:
Inclusion Criteria:

1. Age 12 to < 72 months
2. Refractive error between +3.00D and +6.00D SE (by cycloplegic refraction) in either eye
3. Astigmatism < 1.50D in both eyes
4. Spherical equivalent anisometropia ≤ +1.50D
5. For children 36 to <72 months of age:

   1. No evidence of subnormal visual acuity - Uncorrected monocular visual acuity in both eyes of 20/50 or better for age 36 to <48 months,20/40 or better for age 48 to <60 months, and 20/32 or better for ages 60 to <72 months measured without cycloplegia using the ATS-HOTV© visual acuity testing protocol
   2. Zero (0) or 1 logMAR line interocular difference (IOD) in uncorrected visual acuity measured without cycloplegia using the ATS-HOTV© visual acuity testing protocol
   3. Age-normal stereoacuity on the Randot Preschool Stereotest (see Table 2 of protocol)
6. Gestational age >32 weeks
7. Investigator is willing to prescribe glasses per protocol or observe the hyperopia untreated for 3 years unless specific criteria for deterioration outlined in section 3.3.3 are confirmed.
8. Parent understands the protocol and is willing to accept randomization to either glasses or no glasses initially, and is willing to wear glasses as prescribed or accept that glasses will not be prescribed by the investigator unless specific deterioration criteria outlined in section 3.3.3 are confirmed.
9. Parent has phone (or access to phone) and is willing to be contacted by Jaeb Center staff.
10. Relocation outside of area of an active PEDIG site for this study within the next 36 months is not anticipated.

Exclusion Criteria:

A patient is excluded for any of the following reasons:

1. Any measurable heterotropia at distance (3 meters) or at near (1/3 meter) by cover/uncover testing. Note that patients with heterophoria are eligible.
2. Previous documented strabismus (parental report must be confirmed by investigator)
3. Manifest or latent nystagmus evident clinically
4. Previous treatment of refractive error with glasses or contacts unless duration of glasses or contacts wear was one week or less and occurred more than 2 months prior to enrollment.
5. Previous intraocular, refractive, or extraocular muscle surgery
6. Previous amblyopia treatment
7. Previous vergence/accommodative therapy
8. Parental concerns over learning or development
9. Ocular co-morbidity that may reduce visual acuity
10. Symptoms of blur or asthenopia
11. Developmental delay diagnosed by pediatrician or Individualized Education Program (IEP)
12. Known neurological anomalies (e.g. cerebral palsy, Down syndrome)
13. Inability to perform visual acuity ATS-HOTV testing if ≥ 36 months of age

Ages: 12 Months to 71 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 249 (Actual)
Dates: Start 2012-02-23 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marjean Kulp, OD, MS, Study Chair — Jaeb Center for Health Research; David Petersen, MD, Study Chair — Jaeb Center for Health Research
Locations (2):
- United States (2):
  - The Ohio State University College of Optometry, Columbus, Ohio
  - Rocky Mountain Eye Care Associates, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
In accordance with the NIH data sharing policy, a de-identified database is placed in the public domain on the PEDIG public website after the completion of each protocol and publication of the primary manuscript.
Time Frame: Data will be made available after publication of each primary manuscript.
Access Criteria: Users accessing the data must enter an email address.

REFERENCES:
- [Background] Pediatric Eye Disease Investigator Group. Clinical factors associated with moderate hyperopia in preschool children with normal stereopsis and visual acuity. J AAPOS. 2016 Oct;20(5):455-457. doi: 10.1016/j.jaapos.2016.04.012. Epub 2016 Sep 20. PMID 27663627
- [Result] Pediatric Eye Disease Investigator Group; Kulp MT, Holmes JM, Dean TW, Suh DW, Kraker RT, Wallace DK, Petersen DB, Cotter SA, Manny RE, Superstein R, Roberts TL, Avallone JM, Fishman DR, Erzurum SA, Leske DA, Christoff A. A Randomized Clinical Trial of Immediate versus Delayed Glasses for Moderate Hyperopia in 1- and 2-Year-Olds. Ophthalmology. 2019 Jun;126(6):876-887. doi: 10.1016/j.ophtha.2018.12.049. Epub 2019 Jan 4. PMID 30615896
- [Result] Holmes JM, Kulp MT, Dean TW, Suh DW, Kraker RT, Wallace DK, Petersen DB, Cotter SA, Crouch ER, Lorenzana IJ, Ticho BH, Verderber LC, Weise KK; Pediatric Eye Disease Investigator Group. A Randomized Clinical Trial of Immediate Versus Delayed Glasses for Moderate Hyperopia in Children 3 to 5 Years of Age. Am J Ophthalmol. 2019 Dec;208:145-159. doi: 10.1016/j.ajo.2019.06.021. Epub 2019 Jun 28. PMID 31255587

RESULTS

PARTICIPANT FLOW:
Groups:
- Glasses- Older Cohort; Glasses- Younger Cohort: Glasses are prescribed at enrollment and worn per protocol throughout the duration of the study.
  Glasses: For patients in the glasses group, glasses will be prescribed at enrollment with the sphere cut symmetrically by 1.00D and full cylinder correction. If a subject in the observation group has confirmed deterioration, glasses will be prescribed with amount of correction at investigator discretion.
- Observation- Older Cohort; Observation- Younger Cohort: Glasses will not be prescribed unless the patient has confirmation of one or more deterioration criteria as described in the protocol.
  Glasses: For patients in the glasses group, glasses will be prescribed at enrollment with the sphere cut symmetrically by 1.00D and full cylinder correction. If a subject in the observation group has confirmed deterioration, glasses will be prescribed with amount of correction at investigator discretion.
Period: Overall Study
Arm/Group | Glasses- Older Cohort | Observation- Older Cohort | Glasses- Younger Cohort | Observation- Younger Cohort
Started | 61 | 58 | 65 | 65
Completed | 41 | 43 | 53 | 53
Not Completed | 20 | 15 | 12 | 12
Not completed — Lost to Follow-up | 20 | 15 | 12 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Glasses- Older Cohort | Observation- Older Cohort | Glasses- Younger Cohort | Observation- Younger Cohort | Total
Number analyzed (Participants) | 61 | 58 | 65 | 65 | 249
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 61 | 58 | 65 | 65 | 249
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Customized [Count of Participants; unit: Participants]
  1 Year | 0 | 0 | 42 | 42 | 84
  2 Years | 0 | 0 | 23 | 23 | 46
  3 Years | 19 | 20 | 0 | 0 | 39
  4 Years | 31 | 30 | 0 | 0 | 61
  5 Years | 11 | 8 | 0 | 0 | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 32 | 33 | 35 | 138
  Male | 23 | 26 | 32 | 30 | 111
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2 | 0 | 1 | 0 | 3
  Black/African American | 12 | 14 | 2 | 3 | 31
  Hispanic | 13 | 7 | 7 | 8 | 35
  White | 34 | 35 | 53 | 52 | 174
  More than one race | 0 | 1 | 2 | 2 | 5
  Unknown/Not reported | 0 | 1 | 0 | 0 | 1
Family History of Amblyopia [Count of Participants; unit: Participants] — Population: Family history of amblyopia was not available for 2 (3%) participants in glasses group and 3 (5%) in observation group in the Older Cohort.
  Family history of amblyopia was not reported for 3 participants (5%) in glasses group and 2 participants (3%) in observation group in the Younger Cohort.
  Participants
    number analyzed (Participants) | 59 | 55 | 62 | 63 | 239
    (all) | 16 | 17 | 21 | 20 | 74
Family History of Strabismus [Count of Participants; unit: Participants] — Population: Family history of strabismus was not available for 2 (3%) participants in glasses group and 1 (2%) in the observation group in the Older Cohort.
  Family history of strabismus was not reported for 2 participants (3%) in glasses group in the Younger Cohort.
  Participants
    number analyzed (Participants) | 59 | 57 | 63 | 65 | 244
    (all) | 11 | 16 | 26 | 25 | 78
Diagnosis Of ADHD [Count of Participants; unit: Participants] — ADHD: Attention-Deficit/Hyperactivity Disorder
  Participants | 0 | 0 | 0 | 0 | 0
SE Refractive Error: More hyperopic eye [Count of Participants; unit: Participants] — Refractive error is the measurement of the power of the lenses needed to focus light on the retina. This is measured in diopters (D). Spherical Equivalent is a pair of numbers, one for each eye, that gives an estimate of the refractive error in the eyes. Hyperopia is farsightedness, or a type of refractive error in which things are seen more clearly at a distance than at near. This measurement is in the more hyperopic eye, or the eye that sees worse at near than the other eye.
  Participants
    +2.00D to <+3.00D | 0 | 0 | 0 | 0 | 0
    +3.00D to <+4.00D | 37 | 32 | 25 | 20 | 114
    +4.00D to <+5.00D | 16 | 19 | 19 | 27 | 81
    +5.00D to +6.00D | 8 | 7 | 20 | 13 | 48
    +6.00 to +7.00 D | 0 | 0 | 1 | 5 | 6
    +1.00 to <+2.00 D | 0 | 0 | 0 | 0 | 0
SE Refractive Error: More hyperopic eye [Mean (Standard Deviation); unit: diopters (D)] — Refractive error is the measurement of the power of the lenses needed to focus light on the retina. This is measured in diopters (D). Spherical Equivalent is a pair of numbers, one for each eye, that gives an estimate of the refractive error in the eyes. Hyperopia is farsightedness, or a type of refractive error in which things are seen more clearly at a distance than at near. This measurement is in the more hyperopic eye, or the eye that sees worse at near than the other eye.
  diopters (D) | 3.93 (0.71) | 3.94 (0.74) | 4.32 (0.85) | 4.37 (0.87) | 4.15 (0.82)
SE Refractive Error: Less hyperopic eye [Count of Participants; unit: Participants] — Refractive error is the measurement of the power of the lenses needed to focus light on the retina. This is measured in diopters (D). Spherical Equivalent is a pair of numbers, one for each eye, that gives an estimate of the refractive error in the eyes. Hyperopia is farsightedness, or a type of refractive error in which things are seen more clearly at a distance than at near. This measurement is in the less hyperopic eye, or the eye that sees better at near than the other eye.
  Participants
    +1.00 to <+2.00 D | 0 | 0 | 0 | 1 | 1
    +2.00 to <+3.00D | 10 | 10 | 4 | 2 | 26
    +3.00 to <+4.00D | 34 | 30 | 26 | 27 | 117
    +4.00 to <+5.00D | 12 | 13 | 22 | 21 | 68
    +5.00 to <+6.00D | 5 | 5 | 13 | 11 | 34
    +6.00 to <+7.00D | 0 | 0 | 0 | 3 | 3
SE Refractive Error: Less hyperopic eye [Mean (Standard Deviation); unit: diopters (D)] — Refractive error is the measurement of the power of the lenses needed to focus light on the retina. This is measured in diopters (D). Spherical Equivalent is a pair of numbers, one for each eye, that gives an estimate of the refractive error in the eyes. Hyperopia is farsightedness, or a type of refractive error in which things are seen more clearly at a distance than at near. This measurement is in the less hyperopic eye, or the eye that sees better at near than the other eye.
  diopters (D) | 3.60 (0.78) | 3.59 (0.81) | 4.04 (0.85) | 4.07 (0.90) | 3.84 (0.86)
Anisometropia [Count of Participants; unit: Participants] — Anisometropia is when the refractive error between two eyes is different. The difference in spherical equivalent refraction between the eyes is measured in diopters (D).
  Participants
    0.00 to <+0.50 | 42 | 39 | 47 | 46 | 174
    +0.50D to <+1.00D | 16 | 14 | 13 | 12 | 55
    +1.00D to +1.50D | 3 | 5 | 5 | 7 | 20
Anisometropia [Mean (Standard Deviation); unit: diopters (D)] — Anisometropia is when the refractive error between two eyes is different. The difference in spherical equivalent refraction between the eyes is measured in diopters (D).
  diopters (D) | 0.33 (0.36) | 0.34 (0.34) | 0.28 (0.38) | 0.30 (0.39) | 0.31 (0.37)
Astigmatism: More astigmatic eye [Count of Participants; unit: Participants] — Astigmatism is a condition in which the cornea or lens is irregular shaped/curved. The degree of astigmatism is measured in diopters (D). This measurement is in the more astigmatic eye, or the eye with a larger degree of astigmatism.
  Participants
    0.00D to <+0.50D | 29 | 29 | 36 | 29 | 123
    +0.50D to <+1.00D | 23 | 18 | 18 | 19 | 78
    +1.00D to +1.50D | 9 | 11 | 11 | 17 | 48
Astigmatism: More astigmatic eye [Mean (Standard Deviation); unit: diopters (D)] — Astigmatism is a condition in which the cornea or lens is irregular shaped/curved. The degree of astigmatism is measured in diopters (D). This measurement is in the more astigmatic eye, or the eye with a larger degree of astigmatism.
  diopters (D) | 0.45 (0.45) | 0.44 (0.44) | 0.40 (0.48) | 0.49 (0.48) | 0.45 (0.46)
Astigmatism: Less astigmatic eye [Count of Participants; unit: Participants] — Astigmatism is a condition in which the cornea or lens is irregular shaped/curved. The degree of astigmatism is measured in diopters (D). This measurement is in the less astigmatic eye, or the eye with a smaller degree of astigmatism.
  Participants
    0.00D to <+0.50D | 40 | 41 | 41 | 39 | 161
    +0.50D to <+1.00D | 14 | 12 | 17 | 13 | 56
    +1.00D to +1.50D | 7 | 5 | 7 | 13 | 32
Astigmatism: Less astigmatic eye [Mean (Standard Deviation); unit: diopters (D)] — Astigmatism is a condition in which the cornea or lens is irregular shaped/curved. The degree of astigmatism is measured in diopters (D). This measurement is in the less astigmatic eye, or the eye with a smaller degree of astigmatism.
  diopters (D) | 0.32 (0.42) | 0.25 (0.36) | 0.27 (0.38) | 0.37 (0.47) | 0.31 (0.41)
Distance Visual Acuity: Better-seeing Eye [Count of Participants; unit: Participants] — Distance visual acuity is typically measured by testing the smallest letter or object a patient can identify from 20 feet away. This measurement is recorded as a fraction. The numerator is the distance at which the patient is identifying the letter/object, while the denominator is the distance that a person with normal vision could identify that same object. For example, 20/20 vision is considered normal, where a patient can see at 20 feet what is normally seen at 20 feet. This measurement is for the better-seeing eye, or the eye with better visual acuity. Population: This measure was only used as a baseline characteristic for the Older cohort, no data for this characteristic was collected from the younger cohort.
  Participants
    20/16: number analyzed (Participants) | 61 | 58 | 0 | 0 | 119
    20/16 | 5 | 3 |  |  | 8
    20/20: number analyzed (Participants) | 61 | 58 | 0 | 0 | 119
    20/20 | 16 | 18 |  |  | 34
    20/25: number analyzed (Participants) | 61 | 58 | 0 | 0 | 119
    20/25 | 25 | 18 |  |  | 43
    20/32: number analyzed (Participants) | 61 | 58 | 0 | 0 | 119
    20/32 | 9 | 13 |  |  | 22
    20/40: number analyzed (Participants) | 61 | 58 | 0 | 0 | 119
    20/40 | 6 | 6 |  |  | 12
    20/50: number analyzed (Participants) | 61 | 58 | 0 | 0 | 119
    20/50 | 0 | 0 |  |  | 0
Distance Visual Acuity: Better-seeing Eye [Mean (Standard Deviation); unit: logMAR] — Each visual acuity (VA) measure was assigned a logarithm of minimum angle of resolution (logMAR) equivalent, with 20/20 VA equal to 0 logMAR, and each progressively worse VA equal to an additional 0.1 logMAR. For example:
  20/50 = 0.4 logMAR, 20/40 = 0.3 logMAR, 20/32 = 0.2 logMAR, 20/25 = 0.1 logMAR, 20/20 = 0 logMAR, 20/16 = -0.1 logMAR
  Larger logMAR indicates worse visual acuity.
  This measurement is for the better-seeing eye, or the eye with smaller logMAR visual acuity. Population: This measure was only used as a baseline characteristic for the Older cohort, no data for this characteristic was collected from the younger cohort.
  logMAR
    number analyzed (Participants) | 61 | 58 | 0 | 0 | 119
    (all) | 0.09 (0.11) | 0.10 (0.11) |  |  | 0.10 (0.11)
Distance Visual Acuity: Worse-seeing Eye [Count of Participants; unit: Participants] — Distance visual acuity is typically measured by testing the smallest letter or object a patient can identify from 20 feet away. This measurement is recorded as a fraction. The numerator is the distance at which the patient is identifying the letter/object, while the denominator is the distance that a person with normal vision could identify that same object. For example, 20/20 vision is considered normal, where a patient can see at 20 feet what is normally seen at 20 feet. This measurement is for the worse-seeing eye, or the eye with worse visual acuity. Population: This measure was only used as a baseline characteristic for the Older cohort, no data for this characteristic was collected from the younger cohort.
  Participants
    20/16: number analyzed (Participants) | 61 | 58 | 0 | 0 | 119
    20/16 | 2 | 0 |  |  | 2
    20/20: number analyzed (Participants) | 61 | 58 | 0 | 0 | 119
    20/20 | 7 | 7 |  |  | 14
    20/25: number analyzed (Participants) | 61 | 58 | 0 | 0 | 119
    20/25 | 26 | 25 |  |  | 51
    20/32: number analyzed (Participants) | 61 | 58 | 0 | 0 | 119
    20/32 | 15 | 15 |  |  | 30
    20/40: number analyzed (Participants) | 61 | 58 | 0 | 0 | 119
    20/40 | 8 | 9 |  |  | 17
    20/50: number analyzed (Participants) | 61 | 58 | 0 | 0 | 119
    20/50 | 3 | 2 |  |  | 5
Distance Visual Acuity: Worse-seeing Eye [Mean (Standard Deviation); unit: logMAR] — Each visual acuity (VA) measure was assigned a logarithm of minimum angle of resolution (logMAR) equivalent, with 20/20 VA equal to 0 logMAR, and each progressively worse VA equal to an additional 0.1 logMAR. For example:
  20/50 = 0.4 logMAR, 20/40 = 0.3 logMAR, 20/32 = 0.2 logMAR, 20/25 = 0.1 logMAR, 20/20 = 0 logMAR, 20/16 = -0.1 logMAR
  Larger logMAR indicates worse visual acuity.
  This measurement is for the worse-seeing eye, or the eye with larger logMAR. Population: This measure was only used as a baseline characteristic for the Older cohort, no data for this characteristic was collected from the younger cohort.
  logMAR
    number analyzed (Participants) | 61 | 58 | 0 | 0 | 119
    (all) | 0.15 (0.11) | 0.16 (0.10) |  |  | 0.15 (0.11)
Stereoacuity at Near [Count of Participants; unit: Participants] — Stereoacuity scores (seconds of arc) were calculated based on the Randot Preschool stereoacuity test (scores: 800, 400, 200, 100, 60 and 40). Seconds of arc refers to the visual angle that is being measured in order to determine depth perception. Lower scores indicate better stereoacuity. Population: This measure was only used as a baseline characteristic for the Older cohort, no data for this characteristic was collected from the younger cohort.
  Participants
    40: number analyzed (Participants) | 61 | 58 | 0 | 0 | 119
    40 | 9 | 7 |  |  | 16
    60: number analyzed (Participants) | 61 | 58 | 0 | 0 | 119
    60 | 21 | 12 |  |  | 33
    100: number analyzed (Participants) | 61 | 58 | 0 | 0 | 119
    100 | 13 | 15 |  |  | 28
    200: number analyzed (Participants) | 61 | 58 | 0 | 0 | 119
    200 | 12 | 16 |  |  | 28
    400: number analyzed (Participants) | 61 | 58 | 0 | 0 | 119
    400 | 6 | 6 |  |  | 12
    Nil: number analyzed (Participants) | 61 | 58 | 0 | 0 | 119
    Nil | 0 | 1 |  |  | 1
    Failed pretest: number analyzed (Participants) | 61 | 58 | 0 | 0 | 119
    Failed pretest | 0 | 1 |  |  | 1
Stereoacuity at Near [Median (Full Range); unit: seconds of arc (arcsec)] — Measure Description: Stereoacuity scores (seconds of arc) were calculated based on the Randot Preschool stereoacuity test (scores: 800, 400, 200, 100, 60 and 40). Seconds of arc refers to the visual angle that is being measured in order to determine depth perception. Lower scores indicate better stereoacuity. Population: This measure was only used as a baseline characteristic for the Older cohort, no data for this characteristic was collected from the younger cohort.
  seconds of arc (arcsec)
    number analyzed (Participants) | 61 | 58 | 0 | 0 | 119
    (all) | 100 [40 to 400] | 100 [40 to 400] |  |  | 100 [40 to 400]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Confirmation of Failure Criteria
Description: At the 36-month visit, each subject's condition will be classified as either failure or not a failure. The primary analytic approach will be a treatment group comparison of the proportion meeting failure criteria at 36-months using the Fisher's exact test.
  The participant met failure criteria if ANY of the following criteria (except strabismus surgery prior to the 3-year outcome exam) were met during testing at the 3-year examination both with and without trial frames (without prism or bifocal), and the criteria was confirmed by a retest
  1. Any measurable manifest strabismus in primary gaze at distance or at near not correctable with distance refractive correction alone
  2. Strabismus surgery prior to the 36-month exam
  3. Distance VA below age norms in either eye
  4. ≥2 logMAR lines of IOD if VA is 20/25 or worse in the better-seeing eye
  5. ≥3 logMAR lines of IOD if VA is 20/20 or better in the better-seeing eye
  6. Stereoacuity measured at near below age normal values
Time Frame: 36 months after randomization
Population: Overall number is the number of patients who completed the entire study.
Measure: Count of Participants; unit: Participants
Arm/Group | Glasses- Older Cohort | Observation- Older Cohort | Glasses- Younger Cohort | Observation- Younger Cohort
Number analyzed (Participants) | 41 | 43 | 53 | 53
Participants | 5 | 4 | 11 | 18
Statistical Analysis 1: Comparison: Glasses- Older Cohort vs Observation- Older Cohort; Test type: Other; p = 0.72, Barnard's Exact Test; Risk Difference (RD) = 3, 95% CI 2-sided [-12 to 18]
Statistical Analysis 2: Comparison: Glasses- Younger Cohort vs Observation- Younger Cohort; Test type: Other; p = 0.14, Barnard's Exact Test; Risk Difference (RD) = -13, 95% CI 2-sided [-31 to 4]

2. Secondary Outcome: Subgroup Analysis - Race
Description: Treatment effect in subgroups based on baseline factors will be assessed. Outcome failure status at 36 months will be tabulated by subgroup and reviewed for consistency. Total number of patients who experienced failure at 3 years are shown.
Time Frame: 36 months after randomization
Population: Total number that experienced failure, as reported in primary outcome
Measure: Count of Participants; unit: Participants
Arm/Group | Glasses- Older Cohort | Observation- Older Cohort | Glasses- Younger Cohort | Observation- Younger Cohort
Number analyzed (Participants) | 5 | 4 | 11 | 18
Participants
  Race - Non-white | 2 | 1 | 0 | 4
  Race - White | 3 | 3 | 11 | 14

3. Secondary Outcome: Subgroup Analysis - Gender
Description: as for outcome 2
Time Frame: 36 months
Population: Total number that experienced failure, as reported in primary outcome
Measure: Count of Participants; unit: Participants
Arm/Group | Glasses- Older Cohort | Observation- Older Cohort | Glasses- Younger Cohort | Observation- Younger Cohort
Number analyzed (Participants) | 5 | 4 | 11 | 18
Participants
  Gender- Female | 4 | 3 | 4 | 10
  Gender - Male | 1 | 1 | 7 | 8

4. Secondary Outcome: Subgroup Analysis - Family History of Amblyopia
Description: as for outcome 2
Time Frame: 36 months
Population: Total number that experienced failure, as reported in primary outcome
Measure: Count of Participants; unit: Participants
Arm/Group | Glasses- Older Cohort | Observation- Older Cohort | Glasses- Younger Cohort | Observation- Younger Cohort
Number analyzed (Participants) | 5 | 4 | 11 | 18
Participants
  Family History of Amblyopia- Yes | 3 | 0 | 4 | 6
  Family History of Amblyopia- No | 2 | 4 | 7 | 12

5. Secondary Outcome: Subgroup Analysis - Family History of Strabismus
Description: as for outcome 2
Time Frame: 36 months
Population: Total number that experienced failure, as reported in primary outcome
Measure: Count of Participants; unit: Participants
Arm/Group | Glasses- Older Cohort | Observation- Older Cohort | Glasses- Younger Cohort | Observation- Younger Cohort
Number analyzed (Participants) | 5 | 4 | 11 | 18
Participants
  Family History of Strabismus- Yes | 3 | 0 | 5 | 7
  Family History of Strabismus- No | 2 | 4 | 6 | 11

6. Secondary Outcome: Subgroup Analysis - SE Anisometropia
Description: as for outcome 2
Time Frame: 36 months
Population: Total number that experienced failure, as reported in primary outcome
Measure: Count of Participants; unit: Participants
Arm/Group | Glasses- Older Cohort | Observation- Older Cohort | Glasses- Younger Cohort | Observation- Younger Cohort
Number analyzed (Participants) | 5 | 4 | 11 | 18
Participants
  0.00D to <+0.50D | 3 | 4 | 8 | 14
  +0.50D to <+1.00D | 2 | 0 | 2 | 1
  +1.00D to +1.50D | 0 | 0 | 1 | 3

7. Secondary Outcome: Subgroup Analysis - Mean Refractive Error at Enrollment (Diopters)
Description: as for outcome 2
Time Frame: 36 months
Population: Total number that experienced failure, as reported in primary outcome
Measure: Count of Participants; unit: Participants
Arm/Group | Glasses- Older Cohort | Observation- Older Cohort | Glasses- Younger Cohort | Observation- Younger Cohort
Number analyzed (Participants) | 5 | 4 | 11 | 18
Participants
  +2.50D to <+4.00D | 3 | 2 | 2 | 6
  +4.00D to <+5.00D | 1 | 1 | 5 | 7
  +5.00D to +6.00D | 1 | 1 | 4 | 5

8. Secondary Outcome: Deterioration Criteria Met (Prior to 3 Years)
Description: Estimate of Cumulative Deterioration Rate. Proportion of subjects who deteriorated during the course of the study were evaluated. Reasons for deterioration included stereoacuity, strabismus, treatment due to parental concern, and treatment that was prescribed against protocol.
Time Frame: Enrollment to <36 months
Measure: Count of Participants; unit: Participants
Arm/Group | Glasses- Older Cohort | Observation- Older Cohort | Glasses- Younger Cohort | Observation- Younger Cohort
Number analyzed (Participants) | 61 | 58 | 65 | 65
Participants | 16 | 14 | 20 | 36

9. Secondary Outcome: Mean Change in Spherical Equivalent (SE) Refractive Error (Diopters)
Description: Refractive error is the measurement of the power of the lenses needed to focus light on the retina. This is measured in diopters (D). Spherical Equivalent is a pair of numbers, one for each eye, that gives an estimate of the refractive error in the eyes. Hyperopia is farsightedness, or a type of refractive error in which things are seen more clearly at a distance than at near. Myopia is nearsightedness, or refractive error in which things are seen more clearly at near.
  Mean change in SE refractive error is from baseline to 3 years, measured in diopters. Negative values indicate a shift in the myopic direction.
Time Frame: Enrollment to 3 years
Population: Overall number is the total number of patients who completed the 3-year study.
Measure: Mean (95% Confidence Interval); unit: diopters
Arm/Group | Glasses- Older Cohort | Observation- Older Cohort | Glasses- Younger Cohort | Observation- Younger Cohort
Number analyzed (Participants) | 41 | 43 | 53 | 53
diopters
  More Hyperopic Eye | -0.07 [-0.33 to 0.19] | -0.67 [-0.92 to -0.41] | 0.15 [-0.21 to 0.51] | -0.01 [-0.37 to 0.35]
  Less Hyperopic Eye | 0 [-0.26 to 0.26] | -0.58 [-0.84 to -0.33] | 0.30 [-0.05 to 0.64] | 0.08 [-0.27 to 0.42]
Statistical Analysis 1: Comparison: Glasses- Older Cohort vs Observation- Older Cohort; Analysis for the more hyperopic eye, Older Cohort: An analysis of covariance model adjusting for refractive error at enrollment was used to compare mean change in refractive error between treatment groups; Test type: Other; p = 0.002, ANCOVA — Results are considered statistically significant if p<0.01; Mean Difference (Final Values) = 0.60, 99% CI 2-sided [0.11 to 1.09]
Statistical Analysis 2: Comparison: Glasses- Older Cohort vs Observation- Older Cohort; Analysis for the less hyperopic eye, Older Cohort: An analysis of covariance model adjusting for refractive error at enrollment was used to compare mean change in refractive error between treatment groups; Test type: Other; p = 0.002, ANCOVA — Results are considered statistically significant if p<0.01; Mean Difference (Final Values) = 0.58, 99% CI 2-sided [0.10 to 1.06]
Statistical Analysis 3: Comparison: Glasses- Younger Cohort vs Observation- Younger Cohort; Analysis for the more hyperopic eye, Younger Cohort: An analysis of covariance model adjusting for refractive error at enrollment was used to compare mean change in refractive error between treatment groups; Test type: Other; p = 0.53, ANCOVA — Results are considered statistically significant if p≤0.01; Mean Difference (Final Values) = 0.16, 99% CI 2-sided [-0.51 to 0.84]
Statistical Analysis 4: Comparison: Glasses- Younger Cohort vs Observation- Younger Cohort; Analysis for the less hyperopic eye, Younger Cohort: An analysis of covariance model adjusting for refractive error at enrollment was used to compare mean change in refractive error between treatment groups; Test type: Other; p = 0.38, ANCOVA — Results are considered statistically significant if p≤0.01; Mean Difference (Final Values) = 0.22, 99% CI 2-sided [-0.43 to 0.86]

10. Secondary Outcome: Percentage of Participants With Hyperopia Reduction
Description: Percentage of Participants (%) in which hyperopia reduced by 1.00D (diopters) or more over 3 years
Time Frame: Enrollment to 3 years
Population: Overall number is the number of patients that completed the 3-year study in the Older Cohort. This measure was not recorded for Younger Cohort.
Measure: Number; unit: percentage of participants
Arm/Group | Glasses- Older Cohort | Observation- Older Cohort
Number analyzed (Participants) | 41 | 43
percentage of participants
  More Hyperopic Eye | 17 | 42
  Less Hyperopic Eye | 20 | 37
Statistical Analysis 1: Comparison: Glasses- Older Cohort vs Observation- Older Cohort; Analysis for the more hyperopic eye: Barnard's exact test was used to compare proportions between treatment groups; Test type: Other; p = 0.013, Barnard's Exact Test — Results are considered statistically significant if p<0.01; Mean Difference (Final Values) = -25, 99% CI 2-sided [-49 to 1]
Statistical Analysis 2: Comparison: Glasses- Older Cohort vs Observation- Older Cohort; Analysis for the less hyperopic eye: Barnard's exact test was used to compare proportions between treatment groups; Test type: Other; p = 0.08, Barnard's Exact Test — Results are considered statistically significant if p<0.01; Hazard Ratio, log = -18, 99% CI 2-sided [-42 to 8]

11. Secondary Outcome: Best Visual Acuity
Description: A treatment group comparison of the mean maximum visual acuity per subject at the masked 36-month visit (best visual acuity on any test with and without correction) will be performed using a t-test. Evaluated the best of the values reported with and without trial frames, during initial assessment and retest.
  Snellen visual acuity (VA) equivalents were converted to logarithm of minimum angle of resolution (logMAR) equivalents (in parentheses) as follows: 20/16 (-0.1), 20/20 (0), 20/25 (0.1), 20/32 (0.2), 20/40 (0.3), 20/50 (0.4)
  A logMAR value of less than 0 is associated with better than 20/20 vision, while a logMAR value greater than 0 is associated with worse than 20/20 vision.
Time Frame: 36 months after randomization
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Glasses- Older Cohort | Observation- Older Cohort | Glasses- Younger Cohort | Observation- Younger Cohort
Number analyzed (Participants) | 41 | 43 | 53 | 53
logMAR
  Better-seeing Eye | -0.06 (0.06) | -0.07 (0.05) | 0.06 (0.12) | 0.12 (0.13)
  Worse-seeing Eye | -0.03 (0.08) | -0.01 (0.10) | 0.16 (0.23) | 0.23 (0.26)
Statistical Analysis 1: Comparison: Glasses- Older Cohort vs Observation- Older Cohort; Test for Difference in Means in Better-Seeing Eye: Older Cohort An analysis of covariance model, adjusting for age at the 3-year visit and visual acuity at baseline, was used to compare mean visual acuity between treatment groups. Results are considered statistically significant if p<0.01; Test type: Other; p = 0.22, ANCOVA; Mean Difference (Final Values) = 0.01, 99% CI 2-sided [-0.02 to 0.04]
Statistical Analysis 2: Comparison: Glasses- Older Cohort vs Observation- Older Cohort; Test for Difference in Means in Worse-Seeing Eye: Older Cohort An analysis of covariance model, adjusting for age at the 3-year visit and visual acuity at baseline, was used to compare mean visual acuity between treatment groups. Results are considered statistically significant if p<0.01; Test type: Other; p = 0.41, ANCOVA; Mean Difference (Final Values) = -0.02, 99% CI 2-sided [-0.06 to 0.03]
Statistical Analysis 3: Comparison: Glasses- Younger Cohort vs Observation- Younger Cohort; Test for Difference in Means in Better-Seeing Eye: Younger Cohort An analysis of covariance model, adjusting for age at the 3-year visit and visual acuity at baseline, was used to compare mean visual acuity between treatment groups. Results are considered statistically significant if p<0.01; Test type: Other; p = 0.02, ANCOVA; Mean Difference (Final Values) = -0.05, 99% CI 2-sided [-0.12 to 0.01]
Statistical Analysis 4: Comparison: Glasses- Younger Cohort vs Observation- Younger Cohort; Test for Difference in Means in Worse-Seeing Eye: Younger Cohort An analysis of covariance model, adjusting for age at the 3-year visit and visual acuity at baseline, was used to compare mean visual acuity between treatment groups. Results are considered statistically significant if p<0.01; Test type: Other; p = 0.15, ANCOVA; Mean Difference (Final Values) = -0.07, 99% CI 2-sided [-0.19 to 0.05]

12. Secondary Outcome: Failure to Meet Age-Normal VA at Distance
Description: Proportion who failed to meet age-normal VA at distance at 3 years. Participants were classified as failing to meet age-normal visual acuity if, for either eye, distance visual acuity was below age-normal values both with and without trial frames, during initial assessment and re-test.
Time Frame: 36 months
Population: Overall number is the total number of patients who completed the 3-year study.
Measure: Count of Participants; unit: Participants
Arm/Group | Glasses- Older Cohort | Observation- Older Cohort | Glasses- Younger Cohort | Observation- Younger Cohort
Number analyzed (Participants) | 41 | 43 | 53 | 53
Participants | 0 | 1 | 3 | 4
Statistical Analysis 1: Comparison: Glasses- Older Cohort vs Observation- Older Cohort; Barnard's exact test was used to compare proportions between treatment groups; Test type: Other; p = 0.51, Barnard's Exact Test — Results are considered statistically significant if p<0.01; Mean Difference (Final Values) = -2, 99% CI 2-sided [-18 to 13]
Statistical Analysis 2: Comparison: Glasses- Younger Cohort vs Observation- Younger Cohort; Barnard's exact test was used to compare proportions between treatment groups; Test type: Other; p = 0.79, Barnard's Exact Test — Results are considered statistically significant if p<0.01; Mean Difference (Final Values) = -2, 99% CI 2-sided [-18 to 14]

13. Secondary Outcome: Proportion With Amblyopia (at Distance)
Description: A treatment group comparison of the proportion of subjects who developed amblyopia at distance during the course of the study will be performed using the Barnard's exact test.
  Participants were classified as having amblyopia if any of the following criteria were met: 1) the interocular difference was ≥2 logMAR lines of IOD if VA is 20/25 or worse in the better-seeing eye, or 2) the interocular differences was ≥3 logMAR lines of IOD if VA is 20/20 or better in the better-seeing eye. 3) VA less than age normal in each eye (presumed bilateral amblyopia)
Time Frame: 36 months after randomization
Population: Overall number is the total number of patients who completed the 3-year study.
Measure: Count of Participants; unit: Participants
Arm/Group | Glasses- Older Cohort | Observation- Older Cohort | Glasses- Younger Cohort | Observation- Younger Cohort
Number analyzed (Participants) | 41 | 43 | 53 | 53
Participants | 0 | 1 | 7 | 9
Statistical Analysis 1: Comparison: Glasses- Older Cohort vs Observation- Older Cohort; Barnard's exact test was used to compare proportions between treatment groups; Test type: Other; p = 0.51, Barnard's Exact Test — Results are considered statistically significant if p<0.01; Mean Difference (Final Values) = -2, 99% CI 2-sided [-18 to 13]
Statistical Analysis 2: Comparison: Glasses- Younger Cohort vs Observation- Younger Cohort; Barnard's exact test was used to compare proportions between treatment groups; Test type: Other; p = 0.68, Barnard's Exact Test — Results are considered statistically significant if p≤0.01; Mean Difference (Final Values) = -4, 99% CI 2-sided [-24 to 16]

14. Secondary Outcome: Binocular Near Visual Acuity
Description: A treatment group comparison of the mean binocular near visual acuity (logarithm of minimum angle of resolution, or logMAR) at the 36-month outcome exam will be performed. Assessment completed in randomized correction.
  Snellen visual acuity (VA) equivalents were converted to logarithm of minimum angle of resolution (logMAR) equivalents (in parentheses) as follows: 20/16 (-0.1), 20/20 (0), 20/25 (0.1), 20/32 (0.2), 20/40 (0.3), 20/50 (0.4) A logMAR value of less than 0 is associated with better than 20/20 vision, while a logMAR value greater than 0 is associated with worse than 20/20 vision.
Time Frame: 36 months after randomization
Population: Overall number is the total number of patients who completed the 3-year study.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Glasses- Older Cohort | Observation- Older Cohort | Glasses- Younger Cohort | Observation- Younger Cohort
Number analyzed (Participants) | 41 | 43 | 53 | 53
logMAR | 0.01 (0.04) | 0.04 (0.14) | 0.09 (0.11) | 0.12 (0.12)
Statistical Analysis 1: Comparison: Glasses- Older Cohort vs Observation- Older Cohort; An analysis of covariance model, adjusting for age at the 3-year visit and visual acuity at baseline, was used to compare mean visual acuity between treatment groups; Test type: Other; p = 0.21, ANCOVA — Results are considered statistically significant if p<0.01; Mean Difference (Final Values) = -0.04, 99% CI 2-sided [-0.12 to 0.05]
Statistical Analysis 2: Comparison: Glasses- Younger Cohort vs Observation- Younger Cohort; [analysis description as in outcome 14, analysis 1]; Test type: Other; p = 0.25, ANCOVA — Results are considered statistically significant if p≤0.01; Mean Difference (Final Values) = -0.03, 99% CI 2-sided [-0.10 to 0.04]

15. Secondary Outcome: Number of Participants With Strabismus at 3 Years
Description: The number of participants who developed measurable heterotropia was estimated for each treatment group and the proportions were compared using Barnard's exact test.
Time Frame: 36 months after randomization
Population: In the older cohort, one participant had esotropia. In the younger cohort, Three participants in the glasses group and two in the observation group received strabismus surgery prior to the 3-year visit. These participants are included in the table.
Measure: Count of Participants; unit: Participants
Arm/Group | Glasses- Older Cohort | Observation- Older Cohort | Glasses- Younger Cohort | Observation- Younger Cohort
Number analyzed (Participants) | 41 | 43 | 53 | 53
Participants | 0 | 1 | 5 | 5
Statistical Analysis 1: Comparison: Glasses- Older Cohort vs Observation- Older Cohort; Barnard's exact test used to compare proportions between treatment groups; Test type: Other; p = 0.51, Barnard's Exact Test — Results are considered statistically significant if p<0.01; Mean Difference (Final Values) = -2, 99% CI 2-sided [-18 to 13]
Statistical Analysis 2: Comparison: Glasses- Younger Cohort vs Observation- Younger Cohort; Barnard's exact test used to compare proportions between treatment groups; Test type: Other; No p-value, because there was 0% difference; Mean Difference (Final Values) = 0, 99% CI 2-sided [-17 to 17]

16. Secondary Outcome: Mean Stereoacuity
Description: Mean stereoacuity at 3 years was measured in log seconds of arc (log arcsec) (see explanation below). Evaluated the best of the values reported with and without trial frames, during initial assessment and retest.
  Stereoacuity scores (seconds of arc) were calculated based on the Randot Preschool stereoacuity test (scores: 800, 400, 200, 100, 60 and 40). Seconds of arc refers to the visual angle that is being measured in order to determine depth perception. Lower scores indicate better stereoacuity. A logarithm base 10 transformation was used to convert stereoacuity scores to the log scale to calculate descriptive statistics (reported as seconds of arc, or arcsec). Seconds of arc were converted to logarithm of seconds of arc, or log arcsec (in parentheses) as follows: 40 (1.60), 60(1.78), 100 (2.00), 200 (2.30), 400 (2.60), 800 (2.90), Nil (3.20)
Time Frame: 36 months
Population: Overall number is the total number of patients who completed the 3-year study.
Measure: Mean (Standard Deviation); unit: logarithm of seconds of arc (log arcsec)
Arm/Group | Glasses- Older Cohort | Observation- Older Cohort | Glasses- Younger Cohort | Observation- Younger Cohort
Number analyzed (Participants) | 41 | 43 | 53 | 53
logarithm of seconds of arc (log arcsec) | 1.76 (0.20) | 1.75 (0.23) | 2.2 (0.52) | 2.3 (0.55)
Statistical Analysis 1: Comparison: Glasses- Older Cohort vs Observation- Older Cohort; An analysis of covariance model was used to compare mean change in stereoacuity between treatment groups. The analysis controlled for age at the 3-year visit, anisometropia at the most recent visit, and stereoacuity at enrollment; Test type: Other; p = 0.74, ANCOVA — Results are considered statistically significant if p<0.01; Mean Difference (Final Values) = 0.02, 99% CI 2-sided [-0.11 to 0.14]
Statistical Analysis 2: Comparison: Glasses- Younger Cohort vs Observation- Younger Cohort; An analysis of covariance model was used to compare mean change in stereoacuity between treatment groups. The analysis controlled for age at the 3-year visit and anisometropia at the most recent visit; Test type: Other; p = 0.15, ANCOVA; Mean Difference (Final Values) = -0.1, 99% CI 2-sided [-0.4 to 0.1]

17. Secondary Outcome: Failure to Meet Age-Normal Stereoacuity at 3 Years
Description: Proportion who failed to meet age-normal stereoacuity. Participants were classified as failing to meet age-normal stereoacuity if near stereoacuity was below age-normal values both with and without trial frames, during initial assessment and re-test.
Time Frame: 36 months
Population: Overall number is the total number of patients who completed the 3-year study.
Measure: Count of Participants; unit: Participants
Arm/Group | Glasses- Older Cohort | Observation- Older Cohort | Glasses- Younger Cohort | Observation- Younger Cohort
Number analyzed (Participants) | 41 | 43 | 53 | 53
Participants | 5 | 3 | 6 | 16
Statistical Analysis 1: Comparison: Glasses- Older Cohort vs Observation- Older Cohort; Barnard's exact test used to compare proportions between treatment groups; Test type: Other; p = 0.53, Barnard's Exact Test — Results are considered statistically significant if p<0.01; Mean Difference (Final Values) = 5, 99% CI 2-sided [-14 to 26]
Statistical Analysis 2: Comparison: Glasses- Younger Cohort vs Observation- Younger Cohort; Barnard's exact test used to compare proportions between treatment groups; Test type: Other; p = 0.02, Barnard's Exact Test — Results are considered statistically significant if p<0.01; Mean Difference (Final Values) = -19, 99% CI 2-sided [-40 to 2]

ADVERSE EVENTS:
Time Frame: 3 Years (36 months)
Arm/Group | Glasses- Older Cohort | Observation- Older Cohort | Glasses- Younger Cohort | Observation- Younger Cohort
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/43 | 0/53 | 0/53
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/43 | 0/53 | 0/53
Other Adverse Events (participants affected / at risk) | 0/41 | 0/43 | 0/53 | 0/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Informed Consent Form (2013-10-14): https://cdn.clinicaltrials.gov/large-docs/75/NCT01515475/ICF_000.pdf
  • Statistical Analysis Plan (2018-07-25): https://cdn.clinicaltrials.gov/large-docs/75/NCT01515475/SAP_001.pdf
  • Study Protocol (2015-01-28): https://cdn.clinicaltrials.gov/large-docs/75/NCT01515475/Prot_002.pdf